CLINICAL TRIAL: NCT03004417
Title: A Randomised, Double-blind,Placebo Controlled, Repeated Dose, Three-way Crossover Study to Evaluate the Pharmacodynamics, Pharmacokinetics and Safety of Two Doses of CHF6001 DPI in Subjects With Moderate, Severe COPD
Brief Title: Pharmacodynamics, Pharmacokinetics and Safety of Two Doses of CHF6001 DPI in Subjects With Moderate, Severe COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: SGS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-06001AA1-10; 2015-005550-35 (EudraCT Number)
Record Dates: First submitted 2016-12-02; First posted 2016-12-28 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHF 6001 Dose1 (Experimental): CHF6001 via NEXThaler® dry powder inhaler (DPI), b.i.d. for 32 consecutive days.
  Interventions: Drug: CHF 6001 Dose1
- CHF 6001 Dose 2 (Experimental): CHF6001 via NEXThaler® dry powder inhaler (DPI), b.i.d. for 32 consecutive days.
  Interventions: Drug: CHF 6001 Dose2
- Placebo (Placebo Comparator): Matching placebo via NEXThaler® dry powder inhaler (DPI), b.i.d. for 32 consecutive days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CHF 6001 Dose1 — CHF 6001 plus placebo
  Other Names: CHF 6001
  Arms: CHF 6001 Dose1
Drug: CHF 6001 Dose2 — CHF 6001 only (high dose)
  Other Names: CHF 6001
  Arms: CHF 6001 Dose 2
Other: Placebo — Placebo only
  Arms: Placebo

SUMMARY:
Effect of CHF 6001 on biomarkers of inflammation in induced sputum and in blood, on pulmonary function and on symptoms benefits in comparison with placebo.

DETAILED DESCRIPTION:
The purpose of this study is to obtain information on the effects of two doses of CHF6001 on sputum and blood biomarkers of inflammation in subjects with symptomatic COPD with moderate, severe airflow limitation and with chronic bronchitis. The efficacy of the treatment will also be measured using forced oscillometry technique and spirometry. Safety, tolerability and pharmacokinetics will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged ≥40 years
* A female is eligible to enter the study if she is of non-childbearing potential i.e. physiologically incapable of becoming pregnant Women physiologically capable of becoming pregnant (i.e. women of childbearing potential) are eligible to enter the study if they have negative pregnancy test at screening and agree to use one or more of the following highly effective contraceptive measures
* Subjects with an established diagnosis of COPD (according to GOLD guidelines, update 2015) at least 12 months prior to the screening visit
* With a smoking history of at least 10 pack-years [pack-years=number of cigarettes per day x number of years/20]. Current and ex- smokers are eligible. With a BMI in the range of 18-35 Kg/m2 With a post-bronchodilator FEV1 ≥30% and ≤70%
* Subjects must be receiving daily maintenance with triple therapy (ICS plus LABA plus LAMA) at stable dose and dosing regimen, for at least 2 months prior to screening
* With a history of chronic bronchitis defined as chronic cough and sputum production for more than three months per year for two or more years and known as 'spontaneous sputum producer' subject
* Subjects must be symptomatic at screening defined as having a CAT score ≥10
* Subjects must be able to be trained to correctly use the DPI inhalers and They must have a cooperative attitude and ability to perform the required outcome measurements (e.g. spirometry testing, induced sputum...).

Exclusion Criteria:

* Pregnant or lactating female subject
* Subjects with a current diagnosis of asthma
* Subjects with a moderate or severe COPD exacerbation [i.e. resulting in the use of systemic (oral/IV/IM corticosteroids) and/or antibiotics or in hospitalisation] or a lower respiratory tract infection within 6 weeks prior to study entry or during the screening period
* Subjects on maintenance bronchodilators therapy only (LABA alone, LAMA alone, dual LABA/LAMA alone) or maintenance dual therapy only (ICS/LABA or ICS plus LAMA) within 2 months prior to study entry
* Subjects on PDE4 inhibitors (e.g. roflumilast) within 2 months prior to study entry
* Subjects requiring long-term (at least 12 hours daily) oxygen therapy for chronic hypoxemia; participating to a pulmonary rehabilitation programme or completing such a programme within the last 6 weeks prior to study entry
* Subjects with known respiratory disorders other than COPD...
* Subjects have lung cancer or a history of lung cancer or with active cancer or a history of cancer (other than lung) with less than 5 years disease free survival time
* Subjects with a known history of hypersensitivity to beta2-agonist, PDE4 inhibitors or any of the excipients contained in any of the formulations used in the trial
* Subjects with a diagnosis of depression associated with suicidal ideation or behaviour or with a diagnosis of generalised anxiety disorder that in the investigator's opinion would place the patient at risk
* Subjects who have known history of clinically significant cardiovascular conditions such as, but not limited to, unstable or acute ischemic heart disease within one year prior to study entry, NYHA Class III/IV heart failure, known history of sustained and non-sustained cardiac arrhythmias or history of atrial fibrillation diagnosed in the last 6 months prior to study entry and not controlled with therapy rate control strategy
* Subjects who have unstable concurrent disease
* Subjects with clinically significant laboratory abnormalities
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects receiving treatment with any drug known to have a well-defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole) within the previous 3 months prior to the study entry and during the screening period
* Subjects have experienced excessive weight loss recently (which cannot be explained by the natural course of COPD or known background conditions).
* Subjects with a history of alcohol abuse and/or substance/drug abuse within 12 months prior to screening visit
* Subjects having received any other investigational drug within the preceding 30 days (60 days for biologics).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Sputum biomarkers | Change from baseline to end of treatment (mean Day 20, 26 and 32 values) at each period;
  - IL-6, IL-8 (CXCL-8), IL-1β, TNF-α, MIP1β, MCP-1, MyeloPerOxidase (MPO), Neutrophil Elastase (NE), MMP9, Acetyl-proline-glycine-proline (AcPGP), leukotriene B4 (LTB4), eosinophil cationic protein (ECP) and α2-macroglobulin.
Sputum biomarkers | Predose and end of treatment at Day 32 of each period
  Sputum gene expression analysis
Sputum cell count | Change from baseline to end of treatment (mean Day 20, 26 and 32 values) at each period;
  * Total cell count
  * Absolute and percent of neutrophils, eosinophils, macrophages and lymphocytes differential cell count.
Blood Biomarkers | Change from baseline to Day 32 of each period;
  Blood Biomarkers
Blood Biomarkers | Predose and end of treatment at Day 32 of each period
  Blood gene expression analysis
Lung function: Spirometry | Change from baseline to Day 20 Day 26 and 32 of each period
  pre-dose FEV1, FVC and IC
Lung function: Oscillometry | Change from baseline to Day 32 of each period
  R5, R19, R5-R19, X5, EFL index
PK: AUC0-12h,ss | on Day 32 (steady state) of each period.
PK: Cmax | on Day 32 (steady state) of each period.

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — MEU - Manchester - UK
Locations (1):
- Medicines Evaluation Unit Ltd, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Govoni M, Bassi M, Vezzoli S, Lucci G, Emirova A, Nandeuil MA, Petruzzelli S, Jellema GL, Afolabi EK, Colgan B, Leaker B, Kornmann O, Beeh KM, Watz H, Singh D. Sputum and blood transcriptomics characterisation of the inhaled PDE4 inhibitor CHF6001 on top of triple therapy in patients with chronic bronchitis. Respir Res. 2020 Mar 20;21(1):72. doi: 10.1186/s12931-020-1329-y. PMID 32197620
- [Result] Singh D, Beeh KM, Colgan B, Kornmann O, Leaker B, Watz H, Lucci G, Geraci S, Emirova A, Govoni M, Nandeuil MA. Effect of the inhaled PDE4 inhibitor CHF6001 on biomarkers of inflammation in COPD. Respir Res. 2019 Aug 9;20(1):180. doi: 10.1186/s12931-019-1142-7. PMID 31399091
- [Derived] Govoni M, Bassi M, Santoro D, Donegan S, Singh D. Serum IL-8 as a Determinant of Response to Phosphodiesterase-4 Inhibition in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2023 Sep 1;208(5):559-569. doi: 10.1164/rccm.202301-0071OC. PMID 37192443
- [Derived] Singh D, Watz H, Beeh KM, Kornmann O, Leaker B, Colgan B, Lucci G, Emirova A, Nandeuil MA, Santoro D, Balzano D, Govoni M. COPD sputum eosinophils: relationship to blood eosinophils and the effect of inhaled PDE4 inhibition. Eur Respir J. 2020 Aug 6;56(2):2000237. doi: 10.1183/13993003.00237-2020. Print 2020 Aug. PMID 32341106
- See also: Study Record on EU Clinical Trials Register including results — http://www.clinicaltrialsregister.eu/ctr-search/trial/2015-005550-35